CLINICAL TRIAL: NCT01666119
Title: An Open Label Study To Assess The Safety And Tolerability Of BEMA® Buprenorphine NX In Opioid Dependent Subjects (BNX-201)
Brief Title: An Open Label Study To Assess The Safety And Tolerability Of BEMA® Buprenorphine NX In Opioid Dependent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNX-201
Record Dates: First submitted 2012-08-13; First posted 2012-08-16 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Opioid Dependence
Keywords: Opioid dependence; Suboxone; addiction; BEMA Buprenorphine NX; oral transmucosal
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEMA Buprenorphine NX films (Experimental): BEMA Buprenorphine NX films (3.5/0.6 mg and 5.25/0.9 mg buprenorphine/naloxone)will be provided in 3.361 and 5.447 cm2 film sizes, respectively.
  Interventions: Drug: BEMA Buprenorphine NX films

INTERVENTIONS:
Drug: BEMA Buprenorphine NX films — BEMA Buprenorphine NX films (3.5/0.6 mg and 5.25/0.9 mg buprenorphine/naloxone) will be provided in 3.361 and 5.447 cm2 film sizes, respectively.
  Other Names: BNX

SUMMARY:
This is an open label study in opioid dependent subjects maintained on a stabilized dose of Suboxone tablets or films. The purpose is to assess the safety and tolerability of BEMA Buprenorphine NX administered once daily for 12 weeks to opioid dependent subjects stabilized on Suboxone (buprenorphine/naloxone) tablets or films.

Eligible subjects will be converted to an approximately equal dose of BEMA Buprenorphine NX. This dose will be taken throughout the 12-week treatment period with dose adjustments as clinically indicated for either the control of opioid dependence or adverse events (AEs).

DETAILED DESCRIPTION:
This is an open label study in opioid dependent subjects maintained on a stabilized dose of Suboxone tablets or films.

Eligible subjects will be converted to an approximately equal dose of BEMA Buprenorphine NX. This dose will be taken throughout the 12-week treatment period with dose adjustments as clinically indicated for either the control of opioid dependence or adverse events (AEs). Subjects will be monitored for evidence of buccal irritation attributed to the application of the BEMA Buprenorphine NX film and opioid dependence control according to the Clinical Guidelines for the Use of Buprenorphine in the Treatment of Opioid Addiction - A Treatment Improvement Protocol (TIP 40) guidelines for the use of buprenorphine in the management of opioid dependence.

The total duration of participation for each subject will be up to approximately 18 weeks and includes a Screening period (subjects continue to take Suboxone tablets or films), Baseline visit, a 12-week open label treatment period (subjects take BEMA Buprenorphine NX films and at the Day 84 visit, subjects will return to their prior Suboxone treatment), and a Follow-up Visit.

Vital signs, pulse oximetry, opioid withdrawal symptoms, adverse events (AEs), oral examinations, and concomitant medications will be assessed at intervals throughout the study. Clinical laboratory assessments, urine toxicology and buprenorphine testing, and 12-lead electrocardiograms (ECGs) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained at Screening, prior to any study procedure being performed
2. Male or non-pregnant and non-nursing female. A female of childbearing potential is eligible to participate in this study if she is not pregnant, and is using an acceptable method of birth control
3. Subject is aged 18 to 65 years of age, inclusive
4. Diagnosis of opioid dependence per the Diagnostic and Statistical Manual of Mental Disorders - 4th edition (text revision) (DSM-IV-TR) criteria in the past 12 months including physical dependence on opioids and addiction with compulsive use despite harm
5. Currently taking a stable, single daily dose of 16/4 to 32/8 mg Suboxone tablets or films (buprenorphine/naloxone) for at least 30 days
6. Subject is in good general health; with no clinically significant findings on medical history, physical examination, safety laboratory test and ECG in the judgment of the investigator at screening. Serum creatinine, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) values must be within 3-times the upper limit of normal (ULN). Pulse oximetry must be ≥96%, systolic blood pressure ≥110 mmHg, and diastolic blood pressure ≥65 mmHg.

Exclusion Criteria:

1. Hypokalemia, hypomagnesemia, or clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or clinically significant arrhythmias
2. History of Long QT Syndrome, or an immediate family member with this condition
3. Currently taking Class IA antiarrhythmic medications (eg, quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (eg, sotalol, amiodarone, dofetilide)
4. Uncontrolled hypertension defined as systolic blood pressure >170 mmHg and diastolic blood pressure >90 mmHg at Baseline
5. Pulse oximetry ≤93% at Baseline, regardless of cause
6. Clinically significant abnormality on 12-lead ECG, including a QTc interval >490 milliseconds
7. Use of any medication, nutraceutical or herbal product with CYP3A4 inhibition or induction properties within the past 30 days (see Appendix 4 for a list of applicable drugs). This exclusion also extends to grapefruit juice and grapefruit juice-containing products as well as St. John's wort and St. John's wort-containing products (prescription or nonprescription drugs, vitamins, minerals, or dietary/herbal supplements).
8. Diagnosis of moderate to severe hepatic impairment
9. Use of an investigational drug or device within the last 30 days
10. Participation in a previous clinical study of BEMA Buprenorphine NX or BEMA Buprenorphine
11. History of hypersensitivity, allergy, or intolerance to buprenorphine, naloxone, or related drugs
12. Pierced tongue or mouth
13. Any clinically significant abnormality of the buccal mucosa which could impact drug absorption
14. Suicidal risk, as determined by meeting any of the following:

    1. History of suicidal ideation ≤ 3 months prior to Baseline with a score of 4 (intent to act) or 5 (specific plan and intent) on the eC-SSRS
    2. History of suicidal behavior ≤ 1 year prior to Baseline (actual attempt, interrupted attempt, aborted attempt and/or preparatory acts/behavior) on the eC-SSRS
15. A history or current evidence of any clinically significant disorder or any other condition which in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Sullivan, MD, Principal Investigator — Parkway Medical
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - Haleyville, Alabama
  - Jacksonville, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Prairie Village, Kansas
  - Baltimore, Maryland
  - Fall River, Massachusetts
  - Belvidere, New Jersey
  - Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan JG, Webster L. Novel Buccal Film Formulation of Buprenorphine-Naloxone for the Maintenance Treatment of Opioid Dependence: A 12-Week Conversion Study. Clin Ther. 2015 May 1;37(5):1064-75. doi: 10.1016/j.clinthera.2015.02.027. Epub 2015 Mar 29. PMID 25823919

RESULTS

PARTICIPANT FLOW:
Groups:
- BEMA Buprenorphine NX Films: BEMA Buprenorphine/NX films (3.5/0.6, 5.25/0.9, 7/1.2, 10.5/1.8, and 14/2.4 mg).
  BEMA Buprenorphine/NX films (3.5/0.6, 5.25/0.9, 7/1.2, 10.5/1.8, and 14/2.4 mg).
Period: Overall Study
Arm/Group | BEMA Buprenorphine NX Films
Started | 249
Completed | 197
Not Completed | 52
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 7
Not completed — non compliance with study medication, pa | 18
Not completed — Subject experiencing withdrawal symptoms | 5

BASELINE CHARACTERISTICS:
Arm/Group | BEMA Buprenorphine NX Films
Number analyzed (Participants) | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 164
Region of Enrollment [Number; unit: participants]
  United States | 249

OUTCOME MEASURES:

1. Secondary Outcome: Urine Drug Screen
Description: Urine samples collected at screening and baseline to test for the presence of non-prescribed opioids.
Time Frame: 12 weeks
Population: Subjects with at least one urine drug screen test during the treatment period.
Measure: Number; unit: participants
Groups:
- BEMA Buprenorphine/NX Films: BEMA Buprenorphine/NX films (3.5/0.6mg, 5.25/0.9mg, 7.0/1.2mg, 10.5/1.7mg, 14.0/2.3mg)
Arm/Group | BEMA Buprenorphine/NX Films
Number analyzed (Participants) | 249
participants
  Subjects with +-result for non-prescribed opiod | 19
  Number with single positive result | 11
  Number with 2 positive results | 4
  Number with > 2 positive results | 4

2. Primary Outcome: Adverse Events
Description: Adverse events that occur in more than 2 subjects. Among the adverse events that occurred in > 2 subjects, the total number of unique events that were experienced are reported.
Time Frame: 12 weeks
Population: All subjects who received at least 1 dose of study drug.
Measure: Number; unit: adverse events
Arm/Group | BEMA Buprenorphine/NX Films
Number analyzed (Participants) | 249
adverse events | 36

ADVERSE EVENTS:
Arm/Group | BEMA Buprenorphine NX Films
Serious Adverse Events (participants affected / at risk) | 1/249
Other Adverse Events (participants affected / at risk) | 89/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEMA Buprenorphine NX Films (N=249)
osteomyelitis (Infections and infestations) | 1 (1)
suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEMA Buprenorphine NX Films (N=249)
drug withdrawal syndrome (General disorders) | 89 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No